CLINICAL TRIAL: NCT05834764
Title: Evaluating the Efficacy and Safety of Pyrotinib After Adjuvant Anti-HRE2 Therapy in Women With High-risk in Early or Locally Advanced Stage Breast Cancer
Brief Title: Pyrotinib in Women With High-risk in Early Stage Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Liu Xiaoan, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-BC-II-083
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib (Experimental): pyrotinib 400mg orally daily for one year
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib after anti-HER2 therapy（Trastuzumab combined with Pertuzumab or T-DM1）
  Other Names: Pyrotinib maleate

SUMMARY:
ExteNET study explored neratinib prolong anti-HER2 therapy after trastuzumab therapy found that it can improve disease-free survival in patients with lymph nodes positive; In addition, the subgroup of patients with residual tumors after neoadjuvant therapy was found to improve the survival. However, no conclusive conclusions were reached.

However, since the study was carried out early so only trastuzumab treatment was used, it is urgent to carry out research that is more in line with current clinical practice and bring more benefits to patients. To explore whether pyrotinib can further reduce the risk of recurrence from previously diagnosed HER2-positive breast cancer after treatment with trastuzumab and pertuzumab or T-DM1.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study and sign the informed consent form；
2. Female or male patients, aged ≥ 18 years, and ≤75 years;
3. ECOG PS score: 0-1;
4. Patients with HER2+ early or locally advanced breast cancer confirmed by histopathology: HER2-positive is defined by standard of 3+ by immunohistochemical staining (IHC), or 2+ by immunohistochemical staining (IHC) but positive by in situ hybridization (ISH).
5. Stage II through IIIC HER-2 positive breast cancer with node positive disease after surgery.
6. Been treated for early breast cancer with standard of care duration of trastuzumab combined with pertuzumab or T-DM1.
7. Could have been treated neoadjuvantly but have not reached pathologic complete response.

Exclusion Criteria:

1. metastatic disease (Stage IV) or inflammatory breast cancer
2. Previous or current history of malignant neoplasms, except for curatively treated:Basal and squamous cell carcinoma of the skin,Carcinoma in situ of the cervix.
3. Clinically relevant cardiovascular disease:Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110);
4. A history of allergy to the drugs in this study；
5. Unable or unwilling to swallow tablets
6. History of gastrointestinal disease with diarrhea as the major symptom.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-04-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (iDFS) at year 2 | From enrollment until time of events up to 2 years
  Invasive disease-free survival time is defined as the time from date of enrollment until the first disease recurrence or death from any cause.

SECONDARY OUTCOMES:
Disease-free Survival at year 2 (2y-DFS) | From enrollment until time of events up to 2 years
  Disease-free survival time is defined as the time from date of enrollment until the first disease recurrence（including carcinoma in situ）or death from any cause.
Overall Survival (OS) | Enrollment until death due to any cause, up to 10 years
  Randomization to death from any cause
Invasive Disease-free Survival (iDFS) at year 5 | From enrollment until time of events up to 5 years
  Invasive disease-free survival time is defined as the time from date of enrollment until the first disease recurrence or death from any cause.
AEs and SAEs | From the first administration to one months after the last drug administration
  Adverse events and Adverse events and serious adverse events according to CACTE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoan Liu, Professor, Principal Investigator — Jiangsu Province Hospital/ The First Affiliated Hospital of Nanjing Medical University
Locations (1):
- JiangSu Province Hospital/ The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No